CLINICAL TRIAL: NCT02368314
Title: International Multicenter Randomized Double-blind Comparative Clinical Trial of Safety and Efficacy of BCD-080 (JSC BIOCAD, Russia) and Clexan® (Sanofi Aventis France, France) for Deep Vein Thrombosis Prophylaxis at Orthopedic Surgeries
Brief Title: A Safety and Efficacy Study of BCD-080 Compared to Clexan for Deep Vein Thrombosis Prophylaxis at Orthopedic Surgeries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BCD-080-2
Record Dates: First submitted 2015-02-05; First posted 2015-02-23 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-04

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep vein thrombosis; Prophylaxis; Sodium enoxaparin
MeSH Terms: conditions — Venous Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCD-080 (Experimental): Sodium enoxaparine 40 mg (4 000 anti-Xa IU / 0,4 ml) at pre-filled syringe. Administration of BCD-080 30 mg (0,3 ml) every 12 hours during 14 days after surgery for preventing venous thromboembolic complications after surgery.
  Interventions: Drug: Sodium Enoxaparine
- Clexane (Active Comparator): Sodium enoxaparine 40 mg (4 000 anti-Xa IU / 0,4 ml) at pre-filled syringe. Administration of Clexane 30 mg (0,3 ml) every 12 hours during 14 days after surgery for preventing venous thromboembolic complications after surgery/
  Interventions: Drug: Sodium Enoxaparine

INTERVENTIONS:
Drug: Sodium Enoxaparine — 30 mg (0,3 ml), subcutaneously, twice a day (every 12 h).
  Other Names: Clexane (Sodium Enoxaparine); BCD-080 (Sodium Enoxaparine)

SUMMARY:
The purpose of the study is to prove equivalence of efficacy and safety of BCD-080 and Clexan for deep vein thrombosis and embolism prophylaxis at orthopedic surgeries.

DETAILED DESCRIPTION:
The study will include 116 patients who are planned for hip or knee replacement. Patients will randomized in 2 groups. 1-st group will receive BCD-080 at dose 30 mg every 12 hours during 14 days after surgery, 2-d group will receive Clexane at the same dose. Efficacy assessment will include frequency of deep vein thrombosis (DVT) (proximal and/or distal; symptomatic or asymptomatic), symptomatic nonlethal thromboembolia of the pulmonary artery (PATE) and venous thromboembolism death. Safety assessment will include frequency of "big", "small" and other bleedings and frequency of heparin induced thrombocytopenia.The assessment of efficacy and safety parameters will be made during the treatment and follow-up period (till 60 day).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age ≥18 years and age ≤80 years
3. Women body mass 50-110kg, men body mass 57-110 kg inclusive
4. Patients who are planned for hip or knee replacement
5. Willingness of patients of both sexes and their sexual partners with preserved reproductive function to use reliable methods of contraception, starting from screening and up to 4 weeks after the last dose of the studied drug. This requirement does not apply to patients who underwent surgical sterilization. Reliable methods of contraception involves a 1-barrier method combined with one of the following: spermicides/oral contraceptive
6. Ability of the patient, in the opinion of the investigator, to meet the Protocol requirements.

Exclusion Criteria:

1. Hypersensitivity to the components included in the formula of preparation BCD-080 (CJSC BIOCAD) Clexane (Sanofi-Avensis France, France) or medications of the same class
2. Conditions and diseases in which there is a high risk of bleeding: cerebral aneurysm or aortic dissection, hemorrhagic stroke (including in history)
3. Intractable hemorrhage
4. History of documented diseases of blood coagulation (hemophilia A or B, Willebrand disease and other coagulopathies, idiopathic thrombocytopenic purpura, Heparin induced thrombocytopenia associated with thrombosis or without it, thrombohemorrhagic syndrome, etc.) in anamnesis and/or at the moment of examination
5. Gastric or duodenal ulcer or other erosive and ulcerative lesions of gastrointestinal tract
6. Recent ischemic stroke
7. Uncontrolled severe hypertension; that is, all cases of hypertension, in which blood pressure decrease cannot be achieved with the use of combination of 3 antihypertensive drugs, compulsorily including a diuretic, and non-drug methods of correction (salt-free diet, graduated exercise); or if the results of two successive measurements of supine arterial blood pressure with an interval of 15-30 minutes, systolic blood pressure> 180 mm Hg. or diastolic blood pressure> 105 mm Hg
8. Diabetic or hemorrhagic retinopathy
9. Decompensated diabetes mellitus, diabetes mellitus complications
10. Recent delivery (during last 90 days)
11. Bacterial endocarditis (acute or subacute)
12. Pericarditis and pericardial effusion
13. Renal and/or hepatic insufficiency
14. Intrauterine contraception
15. Surgeries or injuries of brain/spinal cord, spine, eyes, and major surgeries and injuries within 90 days prior to randomization)
16. Spinal surgeries or its deformation in history of patients who are planned for epidural/spinal anesthesia
17. Active liver diseases
18. Anamnestic information about alcoholism, addiction or drug abuse over the last year
19. Contraindications to surgeries
20. Hemoglobin <100 g/l
21. Platelet count <100х10*9/l
22. Creatine clearance <30 ml/min
23. Biochemical blood assay indexes: AST/ALT > UNLх3; total bilirubin > UNLх1,5 (unless other causal factors provided, such as Gilbert's syndrome)
24. Necessity for continued treatment with anticoagulants (except for planned under this study), antiaggregant and fibrinolytics (eg, patients with artificial cardiac valve, atrial fibrillation patients receiving warfarin, etc.)
25. The use of dextrans or fibrinolytic therapy or other drugs affecting hemostasis;
26. Necessity for use of systemic glucocorticosteroids and non-steroidal anti-inflammatory drugs (except for the use of the latter with the purpose of anaesthesia in the early postoperative period - during 3 days after the planned hip or knee replacement)
27. Impossibility of contrast venography: contrast allergy, inability to install an intravenous catheter, etc
28. Pregnancy, lactation period
29. Donation of 450 ml or more of blood or plasma within 60 calendar days before inclusion enrolment
30. Participation in clinical trials no less than 30 days before enrolment into this study or previous participation in this clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashot Agahanyan, MD, Principal Investigator — Railroad Clinical Hospital at the station Chelyabinsk, Chelyabinsk, Russia; Pavel Andreev, MD, PhD, Principal Investigator — Railroad Clinical Hospital at the station Samara, Samara, Russia; Ildar Ahtyamov, Professor, Principal Investigator — State budget institution of further education "Kazan State Medical Academy" the Ministry of Health of the Russian Federation; Valery Zagrekov, MD, PhD, Principal Investigator — Nizhny Novgorod Research Institute of Traumatology and Orthopedics of Public Health Ministry of Russian Federation; Maxim Lucenko, MD, Principal Investigator — Treatment and rehabilitation center of Public Health Ministry of Russian Federation, Moscow; Alexander Sitnik, MD, PhD, Principal Investigator — State Institution "Republican Scientific and Practical Centre for Traumatology and Orthopedics" of the Ministry of Health of the Republic of Belarus
Locations (1):
- Railroad Clinical Hospital at the station Chelyabinsk, Chelyabinsk, Russia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BCD-080 | Clexane
Started | 64 | 60
Completed | 61 | 57
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Population: Population for analysis of safety: all patient who received at least 1 study drug injection.
Groups:
- Total: Total of all reporting groups
Arm/Group | BCD-080 | Clexane | Total
Number analyzed (Participants) | 64 | 59 | 123
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57.50 [53.00 to 63.50] | 60.00 [53.00 to 65.00] | 58.00 [53.00 to 64.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 29 | 24 | 53

OUTCOME MEASURES:

1. Primary Outcome: Frequency of DVT.
Description: Frequency of deep vein thrombosis (DVT) (proximal and/or distal; symptomatic or asymptomatic).
Time Frame: During the treatment period (14 days)
Population: Patient who finished the study as per protocol and had contrast venography results for efficacy evaluation.
Measure: Number; unit: participants
Arm/Group | BCD-080 | Clexane
Number analyzed (Participants) | 59 | 54
participants | 0 | 2
Statistical Analysis 1: Comparison: BCD-080 vs Clexane; Test type: Superiority or Other; p = 0.226, Fisher Exact

2. Primary Outcome: Frequency of Symptomatic Nonlethal Thromboembolia of the Pulmonary Artery (PATE)
Time Frame: During the treatment period (14 days)
Population: Patient who finished the study as per protocol and had contrast venography results for efficacy evaluation.
Measure: Number; unit: participants
Arm/Group | BCD-080 | Clexane
Number analyzed (Participants) | 59 | 54
participants | 0 | 0

3. Primary Outcome: Frequency of Venous Thromboembolism Death
Time Frame: During the treatment period (14 days)
Population: Patient who finished the study as per protocol and had contrast venography results for efficacy evaluation.
Measure: Number; unit: participants
Arm/Group | BCD-080 | Clexane
Number analyzed (Participants) | 59 | 54
participants | 0 | 0

4. Secondary Outcome: Frequency of DTV
Description: Frequency of DTV (proximal and/or distal; symptomatic or asymptomatic)
Time Frame: During the treatment period (14 days) and follow-up period (till 60-th day)
Reporting Status: Not Posted

5. Secondary Outcome: Frequency of Proximal DVT
Description: Frequency of proximal DVT (symptomatic or asymptomatic)
Time Frame: During the treatment period (14 days) and follow-up period (till 60-th day)
Reporting Status: Not Posted

6. Secondary Outcome: Frequency of Distal DVT
Description: Frequency of distal DVT (symptomatic or asymptomatic)
Time Frame: During the treatment period (14 days) and follow-up period (till 60-th day)
Reporting Status: Not Posted

7. Secondary Outcome: Frequency of Symptomatic Nonlethal PATE
Time Frame: During the treatment period (14 days) and follow-up period (till 60-th day)
Reporting Status: Not Posted

8. Secondary Outcome: Frequency of Venous Thromboembolism Death
Time Frame: During the treatment period (14 days) and follow-up period (till 60-th day)
Reporting Status: Not Posted

9. Secondary Outcome: Frequency of Death From Other Causes
Time Frame: During the treatment period (14 days) and follow-up period (till 60-th day)
Reporting Status: Not Posted

10. Secondary Outcome: Frequency of Venous Thromboembolism (PATE and/or DTV)
Time Frame: During the treatment period (14 days) and follow-up period (till 60-th day)
Reporting Status: Not Posted

11. Secondary Outcome: Frequency of "Big" and Clinically Significant "Small" Bleedings
Time Frame: During the treatment period (14 days)
Reporting Status: Not Posted

12. Secondary Outcome: Frequency of "Big" Bleedings
Time Frame: During the treatment period (14 days)
Reporting Status: Not Posted

13. Secondary Outcome: Frequency of Clinically Significant "Small" Bleedings
Time Frame: During the treatment period (14 days)
Reporting Status: Not Posted

14. Secondary Outcome: Frequency of Clinically Significant Bleedings
Time Frame: During the treatment period (14 days)
Reporting Status: Not Posted

15. Secondary Outcome: Frequency of Other "Small" Bleedings
Time Frame: During the treatment period (14 days)
Reporting Status: Not Posted

16. Secondary Outcome: Frequency of All Bleedings
Time Frame: During the treatment period (14 days)
Reporting Status: Not Posted

17. Secondary Outcome: Frequency of Heparin Induced Thrombocytopenia
Time Frame: During the treatment period (14 days)
Reporting Status: Not Posted

18. Secondary Outcome: Frequency of Strokes, Myocardial Infarction, Unstable Angina and Cardiovascular Death
Time Frame: During the treatment period (14 days) and follow-up period (till 60-th day)
Reporting Status: Not Posted

19. Secondary Outcome: Frequency of Other AE SAE
Time Frame: During the treatment period (14 days) and follow-up period (till 60-th day)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | BCD-080 | Clexane
Serious Adverse Events (participants affected / at risk) | 2/64 | 5/59
Other Adverse Events (participants affected / at risk) | 53/64 | 56/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BCD-080 (N=64) | Clexane (N=59)
Sepsis (General disorders) | 1 | 0
Infection of surgery wound surface (Infections and infestations) | 1 | 2
Surgery wound dehiscence (Surgical and medical procedures) | 0 | 1
Large trochanter fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Hemorrhagic discharge from surgical wound (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BCD-080 (N=64) | Clexane (N=59)
Oedema of lower limbs (Vascular disorders) | 0 | 3
Arterial hypertension (Vascular disorders) | 11 | 17
Anemia (Blood and lymphatic system disorders) | 40 | 35
Elevated gamma glutamyl tranferase (Hepatobiliary disorders) | 7 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 3
Elevated D-dimer (Blood and lymphatic system disorders) | 23 | 39
Increase of activated partial thromboplastin time (Blood and lymphatic system disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No